CLINICAL TRIAL: NCT07195513
Title: "PRO-CONNECT" Patient-Reported Outcomes to Coordinate Supportive Care for Unmet Needs During Cancer Treatment
Brief Title: Electronic Patient Reporting of Symptoms and Unmet Needs to Connect Patients With Advanced Cancer to Palliative Care Services
Acronym: PRO-CONNECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Cancer Society (ACS) (Unknown)
Responsible Party: Principal Investigator, Tara.L.Kaufmann, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSDG-23-1019130-01 CTPS
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Palliative Care Referral; Advanced Cancer; Palliative Care, Health Services; Metastatic Cancer (Different Solid Tumour Types)
Keywords: ePROs; Patient Reported Outcomes; Palliative Care; Supportive Care; Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Two-arm pilot randomized controlled trial (n=90; 2:1 allocation) comparing an ePRO-directed referral intervention to palliative/supportive care vs. weekly ePRO symptom monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ePRO-Directed Referral Intervention (Experimental): Participants receive: (1) palliative care education from a trained study coordinator; (2) weekly electronic patient-reported outcome (ePRO) symptom monitoring surveys; (3) monthly ePRO palliative care surveys; and (4) navigation to palliative care services when a referral is placed. Severe or persistent patient-reported symptoms or unmet care needs identified through ePROs will trigger an alert to the oncology team with a recommendation for palliative care referral.
  Interventions: Behavioral: ePRO-Directed Referral and Navigation to Palliative/Supportive Care
- ePRO Symptom Monitoring with Usual Palliative Care Referral (Other): Participants complete weekly electronic patient-reported outcome (ePRO) symptom monitoring surveys as standard care in oncology practice. ePRO results are shared with their oncology team for routine care. Referral to palliative care occurs according to usual clinical practice.
  Interventions: Other: ePRO Symptom Monitoring with Usual Palliative Care Referral

INTERVENTIONS:
Behavioral: ePRO-Directed Referral and Navigation to Palliative/Supportive Care — This intervention combines routine electronic patient-reported outcome (ePRO) symptom monitoring with additional components designed to connect patients more directly to palliative/supportive care. In addition to weekly ePRO symptom surveys, participants complete a monthly palliative care-focused ePRO survey, receive structured palliative care education from a trained study coordinator, and are offered navigation support to facilitate access to palliative/supportive care services. Severe or persistent symptoms or unmet needs reported on ePROs generate an alert to the oncology team along with a recommendation for palliative care referral. This multicomponent approach is intended to address gaps in timely referral and access to palliative/supportive care that are not addressed through symptom monitoring alone.
  Arms: ePRO-Directed Referral Intervention
Other: ePRO Symptom Monitoring with Usual Palliative Care Referral — Participants complete weekly electronic patient-reported outcome (ePRO) symptom monitoring surveys. Survey results are shared with the oncology team to support routine care. Referral to palliative/supportive care is made according to usual clinical practice at the discretion of the oncology team. Unlike the intervention arm, participants do not receive structured palliative care education, a monthly palliative care-focused ePRO survey, navigation support, or referral alerts generated from persistent or severe symptoms and unmet care needs.
  Arms: ePRO Symptom Monitoring with Usual Palliative Care Referral

SUMMARY:
This study is testing whether electronic surveys can help patients with advanced cancer report their symptoms and care needs so their doctors can connect them to palliative/supportive care services sooner. The goal is to see if this approach can make it easier for patients to get support for symptoms, quality of life, and other needs during cancer treatment.

DETAILED DESCRIPTION:
Patients with advanced cancer often experience a range of symptoms and needs while undergoing treatment. Palliative care services aim to address these needs and improve quality of life by preventing and relieving physical, emotional, social, and spiritual suffering.

Palliative care is a specialized type of medical care provided by a team of doctors, nurses, and other professionals who work together with the oncology team. The focus of palliative care is to improve comfort and well-being by treating symptoms such as pain, fatigue, or shortness of breath, and by supporting patients and their families as they cope with the challenges of serious illness. Research has shown that when palliative care is introduced early, patients may experience better symptom control, improved mood and quality of life, and family members may feel less distressed.

Despite these benefits, many patients do not receive timely palliative care because it can be difficult to identify those with unmet needs, and there are not enough specialists available to meet demand.

This study will test a structured approach that uses electronic patient-reported outcomes (ePROs) to support timely referral to palliative care services. Participants in the intervention arm will receive palliative care education from a trained study coordinator, complete weekly ePRO symptom monitoring surveys, and complete monthly ePRO surveys focused on broader palliative care needs. Severe or persistent symptoms reported through these surveys will trigger an alert to the oncology team with a recommendation for palliative care referral. In addition, participants will be offered navigation support to connect with palliative care services.

Participants in the control arm will complete weekly ePRO symptom monitoring surveys, with referral to palliative care occurring according to usual clinical practice.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years.
2. Diagnosis of unresectable or metastatic, incurable thoracic, gastrointestinal, or breast solid tumor.
3. Receiving active cancer-directed therapy longitudinally in the outpatient oncology clinic and expected to continue treatment.

Exclusion Criteria

1. Members of vulnerable populations, including infants, minors, individuals unable to provide informed consent, and those who are incarcerated or imprisoned at the time of enrollment.
2. Already established with palliative care, defined as having a scheduled future palliative care appointment, a pending referral, or a visit with palliative care within the past 90 days.
3. Unable to provide informed consent in English.
4. Cognitive impairment that, in the judgment of the treating clinician, would preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention & Trial Methods | 12 and 24 weeks
  Feasibility will be assessed as a composite of three prespecified components, each summarized as a proportion with 95% confidence intervals:
  Enrollment: Proportion of eligible patients who provide informed consent and are randomized.
  Retention: Proportion of randomized patients who complete the FACT-G at 12 weeks [primary feasibility outcome] and 24 weeks.
  Intervention Compliance:
  Weekly ePRO symptom surveys: Longitudinal compliance quantified as the proportion of participants who self-report at least once in each week of enrollment, averaged over the observation period.
  Monthly palliative-care ePRO surveys (intervention arm): Longitudinal compliance quantified as the proportion of participants who self-report at least once in each month of enrollment, averaged over the observation period.

SECONDARY OUTCOMES:
Referral Rates to Palliative/Supportive Care | 12 and 24 weeks
  Proportion of patients referred to palliative/supportive care during the study period.
Patient Engagement with Palliative Care | 12 and 24 weeks
  Proportion of patients who attend the first palliative care visit among population referred to Palliative Care.
Sustainability | 24 weeks [Exit Survey] / 36 weeks [Study End interviews]
  Recommendation for continued use of the intervention beyond the study period among patients and providers as determined by an Exit Survey and Study End Interview.
Fidelity | From enrollment though end of study at week 24
  Proportion of ePROs delivered to patients, referral alerts sent for ePRO threshold triggers, and patients contacted for palliative care referrals.
Adoption | 12 and 24 weeks
  Proportion of PRO reports and referral alerts viewed by providers.
Appropriateness | 24 weeks [Exit Survey] / 36 weeks [Study End interviews]
  Perceived relevance, usefulness, practicability of the intervention among patients and providers, using an Exit Survey and Study End interview.
Acceptability | 24 weeks [Exit Survey] / 36 weeks [Study End interviews]
  Satisfaction with intervention (content, complexity, comfort, delivery) among patients and providers, using an Exit Survey and optional Study End Interviews.
Health-related Quality of Life | 12 and 24 weeks
  Quality of life as measured by the Functional Assessment of Cancer Therapy-General (FACT-G). Range 0-108 with higher scores indicating better quality of life.
Patient-Reported Pain | 12 and 24 weeks
  Patient-reported pain as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity survey instrument.
  Each question is scored from 1 to 5, where the overall raw survey score ranges from 3-15 with higher scores indicating worse pain.
Patient-reported Mood | 12 and 24 weeks
  Patient-reported mood as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety and Depression survey instruments.
  Each question is scored from 1 to 5 with higher scores indicating more emotional distress (anxiety or depression). For both instruments, the total raw score ranges from 8-40.

OTHER OUTCOMES:
Patient-Centered Communication | 12 and 24 weeks
  Patient-Centered Communication as measured by the Patient-Centered Communication-Cancer-6 (PCC-Ca-6) survey.
  The overall score is a computed average across all completed responses, where the individual responses are scored from 1-5 with higher scores indicating better communication.
Coping Self-Efficacy | 12 and 24 weeks
  Coping self-efficacy as measured by the Cancer Behavior Inventory - Brief Version (CBI-B) survey instrument Individual responses are scored from 1-9, where the total raw score is the sum of all the scored responses, with higher scores indicating better coping abilities.
Aggressive End-Of-Life Care | From enrollment through death (assessed up to 24 weeks)
  Among participants who die during follow-up, proportion meeting any of the following indicators of aggressive end-of-life care: (a) hospice enrollment ≤3 days before death; (b) ≥1 hospitalization within 30 days of death; (c) receipt of chemotherapy within 14 days of death. Components will also be reported separately.
Place of Death Concordance with Preference | From enrollment through death (assessed up to 24 weeks)
  Among participants who die during follow-up, the proportion whose actual place of death matches their documented preferred place of death. Patient preferences will be collected from the electronic health record (EHR).
Advanced Care Planning | Enrollment through 24 weeks
  Proportion of participants with documentation in the electronic health record (EHR) of end-of-life care discussions, such as goals-of-care conversations, preferences for life-sustaining treatment, or hospice discussions, during the study period.
Healthcare Utilization: Emergency Room Visits and Hospitalizations | 12 and 24 weeks
  Average number of emergency room visits and hospitalizations per participant. Data will be collected from the electronic health record (EHR) and from patient surveys. Aggregation method: mean number of visits per participant, with standard deviation (SD), and proportion of participants with ≥1 event at each time point.
Outpatient Palliative Care Utilization | 12 and 24 weeks
  Average number of palliative care visits per participant. Aggregation method: mean number of visits per participant, with standard deviation (SD), and proportion of participants with ≥1 visit at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Tara L. Kaufmann, MD, MSCE, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a small, single-site pilot study of patients with advanced cancer, and the risk of re-identification is high. Preparing de-identified datasets for external use is not feasible for this study.
  Aggregate study results, including feasibility and implementation outcomes, will be shared publicly through ClinicalTrials.gov and peer-reviewed publications. Study protocol and summary materials will be available upon request.

REFERENCES:
- [Background] Kaufmann TL, Kearney M, Cortez D, Saxton JW, Goodfellow K, Smith C, Chang P, Sebastian K, Galaznik A, Scott J, Kvale EA, Kamal AH, Bennett AV, Stover AM, Henneghan AM, Pignone M, Rocque GB. Feasibility Study of Using Electronic Patient-Reported Outcomes to Screen Patients with Advanced Solid Cancers for Palliative Care Needs. J Palliat Med. 2025 May;28(5):580-591. doi: 10.1089/jpm.2024.0375. Epub 2025 Mar 10. PMID 40059654